CLINICAL TRIAL: NCT05062798
Title: The Effect of the Usage of Squeezable vs Standard Bottles on the Feeding Process of Infants With Cleft Lip and Palate (CLP) After Cleft Palate Surgery
Brief Title: The Effect of the Usage of Squeezable vs Standard Bottles After Cleft Palate Surgery on the Feeding Process of Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Zehra Kan Onturk, Assist. Prof., Acibadem University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ATADEK-2021/14
Record Dates: First submitted 2021-09-21; First posted 2021-09-30 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Bottle Feeding
Keywords: infant; cleft lip and palate; Feeding
MeSH Terms: conditions — Bottle Feeding; Cleft Lip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (standart bottle) (Experimental): After the surgery, standard bottle will be used for feeding
  Interventions: Procedure: Standart bottle
- Experimental Group (squeezable bottle) (Experimental): After the surgery, squeezable bottle will be used for feeding
  Interventions: Procedure: Squeezable bottle

INTERVENTIONS:
Procedure: Standart bottle — 1. After the surgery, standard bottle will be used for feeding.
  2. Following the completion of the surgery,feeding process evaluation will be performed until the discharge by using the feeding evaluation form.
  3. Patients will be given a follow-up appointment 2 weeks after the operation and a feeding process evaluation will be made.
  Arms: Control group (standart bottle)
Procedure: Squeezable bottle — 1. After the surgery, squeezable bottle will be used for feeding.
  2. Following the completion of the surgery,feeding process evaluation will be performed until the discharge by using the feeding evaluation form.
  3. Patients will be given a follow-up appointment 2 weeks after the operation and a feeding process evaluation will be made.
  Arms: Experimental Group (squeezable bottle)

SUMMARY:
This study aims to examine the effect of the usage of squeezable bottles and standard bottles on the feeding process of infants with CLP after cleft palate surgery.

DETAILED DESCRIPTION:
Infants with cleft palate commonly have feeding difficulties due to incomplete development of orofacial structures. It has been reported that 67% of infants with cleft palate have feeding difficulties and 86% cannot be breastfed. Feeding difficulties in an infants with a cleft palate can lead to poor weight gain and growth retardation. Therefore, it is essential to provide nutritional interventions for these infants.

This study was designed as a randomized controlled prospective study and was planned to be carried out in the surgical inpatient wards of a private hospital in Istanbul.

Following the diagnosis of cleft lip and palate given to their infants, the families of infants with CLP apply to Aesthetic, Plastic and Reconstructive Surgery Department. In conclusion of the consultations performed in polyclinics, surgery dates are scheduled by the specialist and hospitalization is performed on Surgery Service Ward. Operations of the patients take approximately 3 to 4 hours. Following the operation, for follow-up purposes the patients are taken to Recovery Unit and are observed for 30 to 45 minutes before infants get transferred to Surgical Service. Following the completion of patients' observations in Surgical Service and their transition to full oral feeding, the patients are planned for discharge. The infants continue to be provided with hydration by intravenous infusion until their complete transition to full oral feeding. İnfants with CLP are provided with different nutrition methods before and after surgery. Since the literature also lacks a single or appropriate method that can remove nutrition issues of the babies with CLP, the same nutrition protocol is maintained with an approach in context of resuming the on-going nutrition method after surgery, just like the method previously used before the surgery.

In this study, the patients who use standard bottle before surgery will be included to control group, those who use squeezable bottle will be included to experimental group and participants both will be fed with same methods after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Infants between ≥ 6 to 12 ≤ months,
* Infants with lip, cleft palate and isolated cleft palate anomaly,
* Infants who are being fed using squeezable bottle or standard bottle,
* Infants not having any congenital anomalies or chronic diseases other than CLP,
* Infants with CLP who will undergo CLP surgery,
* Infants who will undergo Cleft Palate surgery

Exclusion Criteria:

* Infants having congenital anomalies or chronic diseases apart from CLP
* Infants who are being fed with a different method rather than using squeezable nipple bottle or standard bottle.

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in oral feed intake | From baseline to transition to total oral feeding (avarege 2 days)
  Change in feed intake will be assessed from baseline to transition to total oral feeding
Change in intravenous infusion intake | From baseline to transition to total oral feeding (avarege 2 days)
  Change in intravenous infusion intake will be assessed from baseline to transition to total oral feeding
Change in body weight | 2 weeks
  Participant's body weight will be assessed from baseline to transition to doctor medical appointment after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Zehra Kan Öntürk, Assist Prof, Principal Investigator — Acibadem University
Locations (1):
- Acıbadem Altunizade Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Duarte GA, Ramos RB, Cardoso MC. Feeding methods for children with cleft lip and/or palate: a systematic review. Braz J Otorhinolaryngol. 2016 Sep-Oct;82(5):602-9. doi: 10.1016/j.bjorl.2015.10.020. Epub 2016 Mar 2. PMID 26997574
- [Result] Farronato G, Cannalire P, Martinelli G, Tubertini I, Giannini L, Galbiati G, Maspero C. Cleft lip and/or palate: review. Minerva Stomatol. 2014 Apr;63(4):111-26. English, Italian. PMID 24705041
- [Result] Miller CK. Feeding issues and interventions in infants and children with clefts and craniofacial syndromes. Semin Speech Lang. 2011 May;32(2):115-26. doi: 10.1055/s-0031-1277714. Epub 2011 Sep 26. PMID 21948638
- [Result] Kumar Jindal M, Khan SY. How to feed cleft patient? Int J Clin Pediatr Dent. 2013 May;6(2):100-3. doi: 10.5005/jp-journals-10005-1198. Epub 2013 Aug 26. PMID 25206201
- [Result] Bessell A, Hooper L, Shaw WC, Reilly S, Reid J, Glenny AM. Feeding interventions for growth and development in infants with cleft lip, cleft palate or cleft lip and palate. Cochrane Database Syst Rev. 2011 Feb 16;2011(2):CD003315. doi: 10.1002/14651858.CD003315.pub3. PMID 21328261